CLINICAL TRIAL: NCT02556138
Title: Endoscopic Intragastric Balloon Placement for Weight Loss in Liver Transplant Waitlist Candidates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain a timely newly requested IDE
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kymberly D. Watt, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-003183
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Obesity; Liver Cirrhosis
Keywords: Intragastric Balloon; ORBERA Intragastric Balloon; Weight Loss; BMI >35
MeSH Terms: conditions — Obesity; Liver Cirrhosis; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Orbera Intragastric Balloon (Experimental): All subjects will be receiving the ORBERA Intragastric Balloon
  Interventions: Device: ORBERA Intragastric Balloon

INTERVENTIONS:
Device: ORBERA Intragastric Balloon — The ORBERA Intragastric Balloon will be placed in the stomach endoscopically through a catheter under conscious sedation. The procedure takes about 20 minutes to complete. The balloon will stay in place for 6 months and then it will be removed endoscopically.

SUMMARY:
The purpose of this study is to determine whether the Orbera Intragastric Balloon is a safe and effective means for weight loss and improved metabolic disease in patients with cirrhosis requiring liver transplantation.

DETAILED DESCRIPTION:
The prevalence of obesity and non-alcoholic steatohepatitis (NASH) in the general population is increasing. More and more patients with underlying NASH-related cirrhosis are now being referred to transplant centers but are not candidates for a potentially lifesaving liver transplantation due to their obesity and comorbidities related to the obesity.

The investigators proposed a clinical pilot study using the new FDA approved intragastric balloon in obese patients (BMI >35) with cirrhosis in need of liver transplantation, to assess weight loss and metabolic improvement.

The ORBERA™ Intragastric Balloon is an elastic spherical balloon made of silicone, filled with 650ml of saline solution. The deflated balloon comes preloaded on a catheter, which is advanced transorally into the stomach. An endoscope is then advanced alongside it to ensure accurate placement of the balloon in the fundus. Under direct visualization, the balloon is then inflated by injecting saline solution mixed with methylene blue through the external portion of the catheter. The ORBERA™ Intragastric Balloon is implanted for 6 months and then retrieved endoscopically by puncturing the balloon with a needle, emptying the fluid content, and removing it through the mouth. Both placement and removal of the ORBERA™ Balloon are done as an outpatient procedure with monitored or general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adults with end-stage liver disease who are listed for liver transplant
* Have failed the non-invasive approach to weight loss to be actively listed for transplant (requiring 2 clinical return visits without weight loss of >5 kg)
* Body Mass Index (BMI) >35
* Negative pregnancy test for females who are able to get pregnant and are of child-bearing age

Exclusion Criteria:

* A previous history of gastric or bariatric surgery
* Current or recent (within 6 months) gastric or duodenal ulcers
* Moderate to severe Portal hypertension defined as portal gastropathy graded as >= to moderate/severe, gastric varices, or esophageal varices graded > = moderate/large (Patients with varices which have been obliterated may be included).
* Calculated Model of End-stage Liver Disease (MELD) score >25 or childs score >10
* The presence of more than one gastric balloon at the same time
* Any inflammatory disease of the gastrointestinal tract including esophagitis, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease.
* A large hiatal hernia or >5 cm hernia or ≤5 cm with associated severe or intractable gastro-esophageal reflux symptoms.
* A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the delivery catheter and/or an endoscope.
* Achalasia or any other severe motility disorder that may pose a safety risk during removal of the device.
* Gastric mass
* Severe coagulopathy
* Patients who are known to have or suspected to have an allergic reaction to materials contained in ORBERA.
* Serious or uncontrolled psychiatric illness or disorder that could compromise patient understanding of or compliance with follow up visits and removal of the device after 6 months.
* Alcoholism or drug addiction
* Patients who are unable or unwilling to take prescribed proton pump inhibitor medication for the duration of the device implant
* Patients unwilling to participate in an established medically-supervised diet and behavior modification program, with routine medical follow-up.
* Patients receiving aspirin, anti-inflammatory agents, anticoagulants or other gastric irritants, not under medical supervision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-11-03 (Actual); Study Completion 2016-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kymberly Watt, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited at the Mayo Clinic in Rochester, Minnesota.
Groups:
- Orbera Intragastric Balloon: All subjects received the ORBERA Intragastric Balloon. The ORBERA Intragastric Balloon was placed in the stomach endoscopically through a catheter under conscious sedation. The procedure took about 20 minutes to complete. The balloon stayed in place for 6 months and then it was removed endoscopically.
Period: Overall Study
Arm/Group | Orbera Intragastric Balloon
Started | 8
Completed | 7 (One patient withdrew from the study due to intolerance of the balloon after 1 month.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Orbera Intragastric Balloon
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With >= 15% Excess Body Weight Loss at 6 Months
Description: The percentage of excess weight loss (%EWL) is a common metric for reporting weight loss after bariatric surgery. The %EWL can vary depending on the definitions of ideal body weight (IBW) used and the preoperative weight.
Time Frame: 6 months
Population: Intent to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Orbera Intragastric Balloon
Number analyzed (Participants) | 8
Participants | 8

2. Secondary Outcome: Mean Percentage of Total Body Weight Loss (%TBWL) After Balloon Removal
Description: %TBWL at 6 months = Number of kg lost at 6 months/starting weight in kg
Time Frame: 6 months
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: percentage of weight loss
Arm/Group | Orbera Intragastric Balloon
Number analyzed (Participants) | 8
percentage of weight loss | 12.3 (8.1)

3. Secondary Outcome: Mean Percentage of Excess Weight Loss (%EWL) After Balloon Removal
Description: as for outcome 1
Time Frame: 6 months
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: percentage of weight loss
Arm/Group | Orbera Intragastric Balloon
Number analyzed (Participants) | 8
percentage of weight loss | 26.3 (16.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Orbera Intragastric Balloon
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orbera Intragastric Balloon (N=8)
Balloon intolerance (Gastrointestinal disorders) | 1 (1)
Liver decompensation (Hepatobiliary disorders) | 2 (2) — balloon retrieved early (1-2 weeks). Liver decompensation was not felt to be due to the balloon.
Mallory-Weiss tears (General disorders) | 2 (2) — Tears due to frequent retching
Hepatocellular carcinoma (Hepatobiliary disorders) | 2 (2)
Retching (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study terminated early as unable to obtain a timely newly requested investigational device exemption (IDE).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes